CLINICAL TRIAL: NCT05865353
Title: Happier Feet- Disrupting the Vicious Cycle of Healthcare Decline in Diabetic Foot Ulceration Through Active Prevention: The Future of Self-managed Care
Brief Title: Happier Feet- A Smart Insole for Diabetic Foot Ulceration Prevention
Acronym: Happier Feet
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: University of Manchester (Other); Loughborough University (Other); University of Southampton (Other); University of Strathclyde (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-22-30; 307041 (Other: IRAS Number)
Record Dates: First submitted 2023-02-06; First posted 2023-05-18 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes: Ten Diabetic participants at risk of DFU/ in this cross-sectional study, participants will be asked to use the smart insole and complete sitting, standing and walking task
- Healthy control: Ten healthy participants without movement disorder or Diabetes. The same tasks (sitting, standing and walking) while wearing the smart insole will be repeated for the control group

SUMMARY:
This study aims to design, develop, and evaluate a smart insole to predict the formation of diabetic foot ulcers (DFUs) in diabetic participants at risk of developing them. The study will be conducted in two phases, using mixed-method research and engaging both diabetic participants and NHS clinicians. In Phase 1, the user-centred design of the smart insole will be developed through focus groups and online questionnaires, and a preliminary safety evaluation of the insole will be conducted with healthy team members. In Phase 2, the insole will be tested, validated, and data will be collected through baseline visits, lab studies, and insole data collection with shape-changed (pressure off-loading) insoles. The study will be conducted by researchers from the University of Manchester and the University of Exeter. It will include 10 people with diabetes and 10 healthy controls in Phase 2.

DETAILED DESCRIPTION:
The tasks in this phase will be conducted by researchers from the University of Manchester and the University of Exeter. All tasks will be held at the University of Exeter.

Recruited participants will attend three sessions (tasks) on three non-consecutive days in the span of three months.

Participants will be identified either through participant identifying centres (e.g., Manchester diabetes clinic) or through direct contact from ad response. From these identified patients, lists will be screened by either general practitioners (for National Health Service (NHS) sites) or the University of Manchester and University o Exeter researchers (for direct contact) according to eligibility criteria. Eligible participants will be written to and invited to return a reply slip detailing whether they are interested in taking part. The return slips will contain all necessary details of the study, including participant information sheets. These must be given to eligible participants at least 48 hours before any planned interview sessions.

Eligible participants that return reply slips, or email the research team to say they are interested, will be contacted by phone by a researcher to clarify any questions they may have. The researcher will then notify the participant of the schedule for the sessions. On the arranged date, before the sessions, the participant will complete the consent process.

n = 20 (10 diabetic participants, 10 healthy similar controls)

1. Task 2.1 Baseline Visit: Eligibility confirmation and health screening session

   * Consented participants will be asked to attend an eligibility confirmation, health evaluation and foot measurements session.
   * This includes:

     * Two-minute walk to evaluate the walking capability
     * Gait and core kinematics evaluation (using IMU sensors and motion capture cameras)
     * Physical Activity Readiness questionnaire (PAR-Q) to determine whether the participant is fit to carry out walking-related activities
     * Monofilament test of the foot (for neuropathy) - Cutaneous pressure perception will be assessed using a 10 g monofilament at the first, third, and fifth prominent metatarsal heads on each foot, with the absence of sensation at any one site indicating neuropathy.
     * Foot measurements and evaluation of anatomical landmarks using a High-Resolution pressure mat (HR-Mat, Tekscan).
     * Participants will also have a fitting session for the co-developed pressure-relief smart insole. Participants will be asked to wear the insoles and give feedback on fitting.

   Data Collection Method:

   - Qualitative data

   Gait and core kinematics evaluation data will be collected in the form of electronic signals (from Intreial Measurement Unit (IMU) sensors) and videos (motion capture cameras)

   Data collected during the baseline visit will be both qualitative and quantitative.
   1. Qualitative data:

      1. Qualitative data may be filled in by the participants at the beginning of the baseline visit or prior to the visit, provided the participants have been given the Participant Information Sheet (PIS) at least 48 hours prior to the visit.
      2. Qualitative data collected within this task are:

      i. Signed participant forms - (i) Decisional capacity evaluation, (ii) consent, (iii) inclusion/exclusion ii. Demographic data - age, sex, weight, iii. Physical Activity Readiness Questionnaire (PAR-Q) iv. Researcher notes v. Monofilament foot test for neuropathy - noted as yes/no for neuropathy.
   2. Quantitative data:

      a. Quantitative data collected within this task are: i. Gait and core kinematics evaluation: using Inertial Measurement Unit (IMU) sensors (physiobiometric) and motion capture cameras and Azure Kinect (data = video files collected and reviewed in the university-managed computer). This will be analysed using Statistical Package for the Social Sciences (SPSS) v.28 or onwards ii. Foot pressure readings (standing) will be collected via HR-Mat in the form of electronic signals that is collected via the HR-Mat Tekscan Research app in a university-managed laptop.
2. Task 2.2 Pilot laboratory - Insole data collection • The first study (Task 2.2) is a pilot evaluation in the lab to collect insole data for a series of activities. The activities are the same between the diabetic and control groups:

   1. Participants will be asked to wear the smart insole while sitting (10 minutes), standing (5 minutes), and walking on a treadmill at a self-selected normal pace (15 minutes).
   2. Participants will be asked to repeat the procedure after a 20 minutes rest.
   3. After repeating the procedure, participants will rest for up to 15 minutes, after which participants will be asked to do a final short 2-5 minute walk on the ground.
   4. Participants will be asked for feedback on the insole and their experience with the study.

      - Participants' health will be monitored throughout the study- heart rate, blood pressure, and blood glucose

      Data Collection Method:

      - Quantitative data Insole data in the form of electronic signals will be collected via the electronic hub (of the insole) and sent via Bluetooth to a university-managed laptop. The data will be recorded and stored in secure folders on the university-managed laptop, followed by further analyses.

      Participant health (heart rate, blood pressure and blood glucose)

      - Qualitative data Qualitative data collected will also be a short questionnaire on the feedback on the usability and acceptability of the insole.

      Participant satisfaction, experience and feedback on the insole/study will be collected through a questionnaire that can either be answered via an electronic questionnaire or a physical copy.
3. Task 2.3 Lab study- insole data collection with shape-changed (pressure shape changed) insole

   * The second study (Task 2.3) pilot evaluation in the lab to collect insole data for a series of activities with a bespoke shape-changed insole to offload the pressures of the foot. The procedures (study methods and data collection) will be as follows:

     1. Participants will be asked to wear the smart insole while sitting (10 minutes), standing (5 minutes), and walking on a treadmill at a self-selected normal pace (15 minutes).
     2. This is followed by a 20-minute rest. During which, a bespoke shape-changed insole will be fitted prior to the next activity.
     3. Participants will repeat #1 with the bespoke shape-changed insole.
     4. After repeating the procedure, participants will rest for up to 15 minutes, after which participants will be asked to do a final short 2-minute walk on the ground.
     5. Participants will be asked for feedback on the insole and their experience with the study.
   * Participants' health will be monitored throughout the study- heart rate, blood pressure, and blood glucose

ELIGIBILITY:
Diabetic Group

Inclusion Criteria:

Confirmed diagnosis of diabetes

1)At the risk of developing a DFU 2) Able to understand and communicate to safely participate [Brief Assessment of Capacity 3) to have a score at least 6/8 (UBACC)]Capacity to participate 4) capability to walk for 10 mins without rest 5) Be able to walk for 30 minutes with no pain, no walking aid, and take breaks if required.

6) Must have sensation on their feet 7) Able to walk without a walking aid or orthotic.

Exclusion Criteria:

1. Below 18 years old
2. Contradictions to walking and physical activity
3. Broken skin on the foot
4. Suffering from a skin condition such as severe eczema or skin allergies
5. Pain affecting the ability to walk.

Healthy participants

Inclusion Criteria:

1. Above 18 years old
2. Able to walk for 30 minutes with no pain, no walking aid, and taking breaks if required.
3. No contraindications to walking and physical activity
4. No broken skin on the foot
5. Do not suffer from a skin condition such as severe eczema or skin allergies.

Exclusion Criteria:

1. below 18 years old
2. Any movement disorder
3. Pain during the walk
4. Broken skin on the foot.
5. suffer from a skin condition such as severe eczema or skin allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises 20 individuals from both genders, divided into two groups: a Diabetic Group consisting of 10 patients with a confirmed diagnosis of diabetes who are at risk of developing or have a history of diabetic foot ulcer (DFU), and a Healthy Control Group consisting of 10 individuals with no diagnosis of diabetes or movement disorder. The selection criteria for the Diabetic Group include a confirmed diagnosis of diabetes and a history or risk of developing DFU, while the Healthy Control Group includes individuals with no known medical conditions that could affect their movement or balance.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Shear data | Participant visit is for 90 minutes and data collection is for the (15 minutes walk, 2 minutes and standing still for 5 minutes)
  Shear data The primary outcome measure includes testing the reliability of the smart insole in collecting
  1. Shear stress data (KPa) while walking at a self-selected speed on the treadmill for 15 minutes
  2. walking on the floor for 2 minutes.
  3. standing on the floor for 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Dawes, PhD, Principal Investigator — Professor of Clinical Rehabilitations; Andrew Weightman, PhD, Principal Investigator — Professor of Medical Mechatronics
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with other researchers or third party